CLINICAL TRIAL: NCT01389856
Title: Multicenter, Double-blind, Placebo-controlled, Randomized, Prospective Study of Bosentan as Adjunctive Therapy to Inhaled Nitric Oxide in the Management of Persistent Pulmonary Hypertension of the Newborn (PPHN)
Brief Title: Persistent Pulmonary Hypertension of the Newborn
Acronym: FUTURE 4
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: To be compliant with the timelines as agreed with Paediatric Committee (PC) within the Paediatric Investigational Plan
Sponsor: Actelion (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: AC-052-391
Record Dates: First submitted 2011-06-30; First posted 2011-07-08 (Estimated); Results first posted 2015-03-23 (Estimated); Last update posted 2025-02-04 (Actual); Status verified 2025-01

CONDITIONS: Persistent Pulmonary Hypertension of the Newborn
Keywords: Persistent pulmonary hypertension, newborn; PPHN
MeSH Terms: conditions — Persistent Fetal Circulation Syndrome | interventions — Bosentan

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): Bosentan
  Interventions: Drug: Bosentan
- 2 (Placebo Comparator): Matching placebo
  Interventions: Drug: Matching placebo

INTERVENTIONS:
Drug: Bosentan — 2 mg/kg of weight at birth twice daily (b.i.d); quadrisectable 32 mg tablet of bosentan dispersed in sterile water and administered by nasogastric or orogastric tube.
  Other Names: Tracleer
  Arms: 1
Drug: Matching placebo — twice daily (b.i.d); quadrisectable 32 mg tablet of matching placebo dispersed in sterile water and administered by nasogastric or orogastric tube.
  Arms: 2

SUMMARY:
The AC-052-391-study is a phase 3 study to investigate whether adding bosentan to inhaled nitric oxide in newborns with persistent pulmonary hypertension of newborns (PPHN) is a supporting and safe therapy and to evaluate the pharmacokinetics of bosentan and its metabolites.

ELIGIBILITY:
Inclusion Criteria:

1. Signed informed consent by the parent(s) or the legal representative(s).
2. Term and near term newborns (gestational age > 34 weeks).
3. Post natal age ≥ 12 hours and < 7 days.
4. Weight at birth ≥ 2,000 g.
5. Idiopathic PPHN or PPHN due to parenchymal lung disease
6. Documented diagnosis of pulmonary hypertension (PH) confirmed by echocardiography.
7. Need for continued inhaled nitric oxide (iNO) at a dose > 10ppm after at least 4 hours of continuous iNO treatment.
8. Two oxygenation index (OI) values ≥ 12 taken at least 30 minutes apart, in the 12 hours prior to randomization and while the patient is receiving iNO treatment.
9. Mechanical ventilation with fraction of inspired oxygen (FiO2) ≥ 50% at randomization.

Exclusion Criteria:

1. PH associated with conditions other than PPHN.
2. Immediate need for cardiac resuscitation or extracorporeal membrane oxygenation (ECMO).
3. Lethal congenital anomalies.
4. Congenital Diaphragmatic Hernia.
5. Significant structural cardiac anomalies.
6. Medically significant pneumothorax.
7. Active seizures.
8. Expected duration of mechanical ventilation of less than 48 hours.
9. Mean systemic blood pressure < 35 mmHg despite therapy with volume infusions and cardiotonic support.
10. Hepatic failure or all conditions with alanine aminotransferase (ALT) values > 2 x upper limit of normal (ULN).
11. Renal function impairment such as serum creatinine > 3 x ULN or anuria.
12. Known intracranial hemorrhage grade III or IV.
13. Either hemoglobin or hematocrit level < 75% of the lower limit of normal (LLN).
14. Thrombocytopenia (platelet count < 50,000 cells /µL).
15. Leukopenia (WBC < 2,500 cells/ µL).
16. Any condition precluding the use of a nasogastric/orogastric tube.
17. Administration of prohibited medication prior to randomization.

Ages: 12 Hours to 7 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 23 (Actual)
Dates: Start 2011-12; Primary Completion 2013-12 (Actual); Study Completion 2014-01 (Actual)

REFERENCES:
- [Derived] Steinhorn RH, Fineman J, Kusic-Pajic A, Cornelisse P, Gehin M, Nowbakht P, Pierce CM, Beghetti M; FUTURE-4 study investigators. Bosentan as Adjunctive Therapy for Persistent Pulmonary Hypertension of the Newborn: Results of the Randomized Multicenter Placebo-Controlled Exploratory Trial. J Pediatr. 2016 Oct;177:90-96.e3. doi: 10.1016/j.jpeds.2016.06.078. Epub 2016 Aug 5. PMID 27502103

RESULTS

PARTICIPANT FLOW:
Recruitment Details: First patient, first visit was 8 December 2011 and last patient, last visit was 5 December 2013. The investigational sites were tertiary care centers with neonatal intensive care unit facilities at which inhaled nitric oxide (iNO) was used as standard of care for persistent pulmonary hypertension of the newborn (PPHN).
Pre-assignment Details: Term or near-term (gestational age > 34 weeks) hypoxic newborns with respiratory distress refractory to supplemental oxygen were considered, provided they had no significant structural cardiac anomalies documented in the pre-natal period and had no immediate need for extra corporeal membrane oxygenation (ECMO).
Groups:
- Bosentan: Bosentan
  Bosentan: 2 mg/kg of weight at birth twice daily (b.i.d); quadrisectable 32 mg tablet of bosentan dispersed in sterile water and administered by nasogastric or orogastric tube.
- Placebo: Matching placebo
  Matching placebo: twice daily (b.i.d); quadrisectable 32 mg tablet of matching placebo dispersed in sterile water and administered by nasogastric or orogastric tube.
Period: Overall Study
Arm/Group | Bosentan | Placebo
Started | 13 (Randomized and treated. An additional 2 patients were randomized but not treated.) | 8 (Randomized and treated.)
Completed | 13 | 8
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Randomized and treated patients
Groups:
- Total: Total of all reporting groups
Arm/Group | Bosentan | Placebo | Total
Number analyzed (Participants) | 13 | 8 | 21
Age, Continuous [Median (Full Range); unit: days] | 1.4 [0.6 to 5.6] | 1.7 [0.6 to 5.9] | 1.4 [0.6 to 5.9]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 6 | 15
  Male | 4 | 2 | 6
Race/Ethnicity, Customized [Number; unit: participants]
  Caucasian/white | 11 | 6 | 17
  Asian | 1 | 0 | 1
  Hispanic | 1 | 1 | 2
  Other | 0 | 1 | 1
Region of Enrollment [Number; unit: participants]
  Czech Republic | 1 | 1 | 2
  France | 1 | 0 | 1
  Korea, Republic of | 1 | 0 | 1
  Poland | 5 | 3 | 8
  United Kingdom | 4 | 2 | 6
  United States | 1 | 2 | 3
Gestational age [Median (Full Range); unit: weeks] | 40.0 [36.0 to 41.0] | 38.5 [36.0 to 42.0] | 39.0 [36.0 to 42.0]

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Patients With Treatment Failure
Description: Treatment failure was defined as the need for extra corporeal membrane oxygenation or initiation of alternative pulmonary vasodilator treatment
Time Frame: From baseline to up to 21 days
Population: Randomized and treated patients
Measure: Number; unit: percentage of participants
Arm/Group | Bosentan | Placebo
Number analyzed (Participants) | 13 | 8
percentage of participants | 7.7 | 0
Statistical Analysis 1: Comparison: Bosentan vs Placebo; Test type: Superiority or Other; p = 1, Fisher Exact

2. Primary Outcome: Time to Complete Weaning From iNO
Description: Calculated from the time from first study drug administration to complete weaning from iNO. Weaning from iNO was considered complete if there was no requirement for the re-initiation of iNO within 24 h after stopping
Time Frame: From baseline to up to 21 days
Population: Randomized and treated patients
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Bosentan | Placebo
Number analyzed (Participants) | 13 | 8
days | 3.7 [1.17 to 6.95] | 2.9 [1.26 to 4.23]
Statistical Analysis 1: Comparison: Bosentan vs Placebo; Test type: Superiority or Other; p = 0.3407, Log Rank

3. Primary Outcome: Time to Complete Weaning From Mechanical Ventilation
Description: Calculated from the time from first study drug administration to complete weaning from mechanical ventilation
Time Frame: From baseline to up to 21 days
Population: Randomized and treated patients
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Bosentan | Placebo
Number analyzed (Participants) | 13 | 8
days | 10.8 [3.21 to 12.21] | 8.6 [3.71 to 9.66]
Statistical Analysis 1: Comparison: Bosentan vs Placebo; Test type: Superiority or Other; p = 0.2399, Log Rank

4. Secondary Outcome: Percentage of Patients Requiring Re-initiation of iNO Therapy
Description: Re-initiation of iNO therapy following weaning from iNO therapy
Time Frame: From baseline to up to 21 days
Population: Randomized and treated patients
Measure: Number; unit: percentage of participants
Arm/Group | Bosentan | Placebo
Number analyzed (Participants) | 13 | 8
percentage of participants | 0 | 0

5. Secondary Outcome: Percentage of Patients With Pulmonary Hypertension (PH) at End of Treatment
Description: The presence of PH was assessed by echocardiography. PH was reported as 'present' if at least one of the following criteria was met:
  * Shunt through ductus arteriosus was either 'predominant right to left' or 'bidirectional'
  * Shunt through foramen ovale was either 'predominant right to left' or 'bidirectional'
  * Marked right ventricular dilation was ticked 'present'
  * Paradoxical shift of intraventricular septum was ticked 'present'
  * Right ventricular systolic pressure (mmHg) was > 2/3 of the reported systemic blood pressure
Time Frame: From baseline to up to 14 days
Population: Randomized and treated patients
Measure: Number; unit: percentage of participants
Arm/Group | Bosentan | Placebo
Number analyzed (Participants) | 13 | 8
percentage of participants | 41.7 | 37.5
Statistical Analysis 1: Comparison: Bosentan vs Placebo; Test type: Superiority or Other; p = 1.000, Fisher Exact

6. Secondary Outcome: Change in Oxygenation Index (OI) From Baseline to 3 Hours Following Study Drug Administration
Description: The change in OI from baseline following study drug administration was determined. OI was calculated as the mean airway pressure multiplied by the fraction of inspired oxygen (expressed in %), and the product was divided by the partial pressure of oxygen in arterial blood.
Time Frame: 3 hours
Population: Randomized and treated patients
Measure: Median (95% Confidence Interval); unit: oxygenation index
Arm/Group | Bosentan | Placebo
Number analyzed (Participants) | 13 | 8
oxygenation index
  Baseline | 18.3 [8.2 to 35.4] | 13.2 [7.9 to 39.4]
  3 hours | 17.3 [6.9 to 33.3] | 13.0 [8.5 to 42.9]
  Change from baseline | -1.6 [-5.1 to 3.3] | 1.1 [-6.1 to 6.1]
Statistical Analysis 1: Comparison: Bosentan vs Placebo; Test type: Superiority or Other; p = 0.2235, Non-parametric ANCOVA

7. Secondary Outcome: Change in Oxygenation Index (OI) From Baseline to 5 Hours Following Study Drug Administration
Description: as for outcome 6
Time Frame: 5 hours
Population: Randomized and treated patients
Measure: Median (95% Confidence Interval); unit: oxygenation index
Arm/Group | Bosentan | Placebo
Number analyzed (Participants) | 13 | 8
oxygenation index
  Baseline | 18.3 [8.2 to 35.4] | 13.2 [7.9 to 39.4]
  5 hours | 16.7 [7.9 to 36.7] | 13.3 [6.7 to 28.6]
  Change from baseline | -0.9 [-4.7 to 4.5] | -5.6 [-7.5 to 15.7]
Statistical Analysis 1: Comparison: Bosentan vs Placebo; Test type: Superiority or Other; p = 0.1468, Non-parametric ANCOVA

8. Secondary Outcome: Change in Oxygenation Index (OI) From Baseline to 12 Hours Following Study Drug Administration
Description: as for outcome 6
Time Frame: 12 hours
Population: Randomized and treated patients
Measure: Median (95% Confidence Interval); unit: oxygenation index
Arm/Group | Bosentan | Placebo
Number analyzed (Participants) | 13 | 8
oxygenation index
  Baseline | 18.3 [8.2 to 35.4] | 13.2 [7.9 to 39.4]
  12 hours | 14.3 [8.3 to 26.7] | 11.1 [4.9 to 19.6]
  Change from baseline | -0.8 [-12.9 to 2.8] | -3.9 [-14.6 to 12.5]
Statistical Analysis 1: Comparison: Bosentan vs Placebo; Test type: Superiority or Other; p = 0.0789, Non-parametric ANCOVA

9. Secondary Outcome: Change in Oxygenation Index (OI) From Baseline to 24 Hours Following Study Drug Administration
Description: as for outcome 6
Time Frame: 24 hours
Population: Randomized and treated patients
Measure: Median (95% Confidence Interval); unit: oxygenation index
Arm/Group | Bosentan | Placebo
Number analyzed (Participants) | 13 | 8
oxygenation index
  Baseline | 18.3 [8.2 to 35.4] | 13.2 [7.9 to 39.4]
  24 hours | 13.1 [6.5 to 32.9] | 11.8 [5.2 to 26.4]
  Change from baseline | -4.9 [-17.0 to 1.1] | -6.9 [-9.9 to 19.4]
Statistical Analysis 1: Comparison: Bosentan vs Placebo; Test type: Superiority or Other; p = 0.3723, Non-parametric ANCOVA

10. Secondary Outcome: Change in Oxygenation Index (OI) From Baseline to 48 Hours Following Study Drug Administration
Description: as for outcome 6
Time Frame: 48 hours
Population: Randomized and treated patients with available data
Measure: Median (95% Confidence Interval); unit: oxygenation index
Arm/Group | Bosentan | Placebo
Number analyzed (Participants) | 12 | 8
oxygenation index
  Baseline | 19.4 [8.2 to 35.4] | 13.2 [7.9 to 39.4]
  48 hours | 11.5 [4.7 to 21.0] | 3.8 [2.5 to 10.8]
  Change from baseline | -4.9 [-15.5 to -2.1] | -9.9 [-18.0 to 3.4]
Statistical Analysis 1: Comparison: Bosentan vs Placebo; Test type: Superiority or Other; p = 0.0569, Non-parametric ANCOVA

11. Secondary Outcome: Change in Oxygenation Index (OI) From Baseline to 72 Hours Following Study Drug Administration
Description: as for outcome 6
Time Frame: 72 hours
Population: Randomized and treated patients with available data
Measure: Median (95% Confidence Interval); unit: oxygenation index
Arm/Group | Bosentan | Placebo
Number analyzed (Participants) | 12 | 8
oxygenation index
  Baseline | 19.4 [8.2 to 35.4] | 13.2 [7.9 to 39.4]
  72 hours | 6.7 [4.2 to 17.0] | 3.9 [3.7 to 10.8]
  Change from baseline | -8.9 [-23.1 to -1.8] | -9.4 [-17.7 to 2.2]
Statistical Analysis 1: Comparison: Bosentan vs Placebo; Test type: Superiority or Other; p = 0.1015, Non-parametric ANCOVA

12. Secondary Outcome: Change in Arterial Blood Gas (ABG) pH From Baseline to 72 Hours Following Study Drug Administration
Description: pH was determined in arterial blood samples at baseline and 72 h after the first study drug administration
Time Frame: 72 hours
Population: Randomized and treated patients with available data
Measure: Median (95% Confidence Interval); unit: pH
Arm/Group | Bosentan | Placebo
Number analyzed (Participants) | 12 | 8
pH
  Baseline | 7.37 [7.30 to 7.43] | 7.31 [7.21 to 7.49]
  72 hours | 7.37 [7.36 to 7.43] | 7.36 [7.30 to 7.39]
  Change from baseline | 0.04 [-0.06 to 0.07] | 0.02 [-0.09 to 0.19]
Statistical Analysis 1: Comparison: Bosentan vs Placebo; Test type: Superiority or Other; p = 0.0824, Non-parametric ANCOVA

13. Secondary Outcome: Change in Arterial Blood Oxygen Saturation (SaO2) From Baseline to 72 Hours Following Study Drug Administration
Description: SaO2 was determined in arterial blood samples at baseline and 72 h after the first study drug administration
Time Frame: 72 hours
Population: Randomized and treated patients with available data
Measure: Median (95% Confidence Interval); unit: percentage saturation
Arm/Group | Bosentan | Placebo
Number analyzed (Participants) | 11 | 8
percentage saturation
  Baseline | 95.0 [92.0 to 99.0] | 95.5 [89.0 to 99.0]
  72 hours | 98.0 [95.0 to 100.0] | 97.0 [93.0 to 100.0]
  Change from baseline | 1.0 [0.0 to 8.0] | 0.0 [-4.0 to 21.0]
Statistical Analysis 1: Comparison: Bosentan vs Placebo; Test type: Superiority or Other; p = 0.3863, Non-parametric ANCOVA

14. Secondary Outcome: Change in Partial Pressure of Oxygen (PaO2) in Arterial Blood From Baseline to 72 Hours Following Study Drug Administration
Description: PaO2 was determined in arterial blood samples at baseline and 72 h after the first study drug administration
Time Frame: 72 hours
Population: Randomized and treated patients with available data
Measure: Median (95% Confidence Interval); unit: mm Hg
Arm/Group | Bosentan | Placebo
Number analyzed (Participants) | 12 | 8
mm Hg
  Baseline | 61.0 [53.0 to 132.0] | 69.5 [46.0 to 111.0]
  72 hours | 81.0 [61.0 to 104.0] | 81.5 [56.0 to 187.0]
  Change from baseline | 18.0 [-13.0 to 32.0] | 6.0 [-12.0 to 115.0]
Statistical Analysis 1: Comparison: Bosentan vs Placebo; Test type: Superiority or Other; p = 0.3936, Non-parametric ANCOVA

15. Secondary Outcome: Change in Partial Pressure of Carbon Dioxide (PaCO2) in Arterial Blood From Baseline to 72 Hours Following Study Drug Administration
Description: PaCO2 was determined in arterial blood samples at baseline and 72 h after the first study drug administration
Time Frame: 72 hours
Population: Randomized and treated patients with available data
Measure: Median (95% Confidence Interval); unit: mm Hg
Arm/Group | Bosentan | Placebo
Number analyzed (Participants) | 12 | 8
mm Hg
  Baseline | 40.5 [31.0 to 47.0] | 46.0 [35.0 to 57.0]
  72 hours | 45.5 [36.0 to 49.0] | 46.0 [41.0 to 64.0]
  Change from baseline | 6.0 [-1.0 to 12.0] | 8.0 [-8.0 to 21.0]
Statistical Analysis 1: Comparison: Bosentan vs Placebo; Test type: Superiority or Other; p = 0.2436, Non-parametric ANCOVA

16. Secondary Outcome: Change in Pre-ductal Peripheral Oxygen Saturation (SpO2) From Baseline to 72 Hours Following Study Drug Administration
Description: Simultaneous pre- (right hand) and post-ductal (lower extremities) SpO2 were measured using pulse oximetry device at baseline and 72 h after the first study drug administration
Time Frame: 72 hours
Population: Randomized and treated patients with available data
Measure: Median (95% Confidence Interval); unit: percentage saturation
Arm/Group | Bosentan | Placebo
Number analyzed (Participants) | 12 | 7
percentage saturation
  Baseline | 95.00 [91.00 to 99.00] | 97.00 [91.00 to 99.00]
  72 hours | 96.00 [93.00 to 100.00] | 96.00 [85.00 to 100.00]
  Change from baseline | 0.50 [-2.00 to 2.00] | -1.00 [-10.00 to 2.00]
Statistical Analysis 1: Comparison: Bosentan vs Placebo; Test type: Superiority or Other; p = 0.1756, Non-parametric ANCOVA

17. Secondary Outcome: Change in Post-ductal Peripheral Oxygen Saturation (SpO2) From Baseline to 72 Hours Following Study Drug Administration
Description: as for outcome 16
Time Frame: 72 hours
Population: Randomized and treated patients with available data
Measure: Median (95% Confidence Interval); unit: percentage saturation
Arm/Group | Bosentan | Placebo
Number analyzed (Participants) | 12 | 8
percentage saturation
  Baseline | 96.5 [92.0 to 99.0] | 96.0 [89.0 to 98.0]
  72 hours | 95.5 [94.0 to 99.0] | 97.5 [95.0 to 100.0]
  Change from baseline | 0.0 [-2.0 to 3.0] | 2.0 [1.0 to 12.0]
Statistical Analysis 1: Comparison: Bosentan vs Placebo; Test type: Superiority or Other; p = 0.1155, Non-parametric ANCOVA

18. Secondary Outcome: Change in Fraction of Inspired Oxygen (FiO2) From Baseline to 72 Hours Following Study Drug Administration
Description: FiO2 was determined according to each study centers' standard procedure at baseline and 72 h after the first study drug administration
Time Frame: 72 hours
Population: Randomized and treated patients with available data
Measure: Median (95% Confidence Interval); unit: percentage of oxygen
Arm/Group | Bosentan | Placebo
Number analyzed (Participants) | 12 | 8
percentage of oxygen
  Baseline | 90.0 [62.0 to 97.0] | 78.0 [60.0 to 100.0]
  72 hours | 51.5 [28.0 to 60.0] | 40.0 [25.0 to 60.0]
  Change from baseline | -33.5 [-50.0 to -15.0] | -35.5 [-60.0 to 0.0]
Statistical Analysis 1: Comparison: Bosentan vs Placebo; Test type: Superiority or Other; p = 0.1400, Non-parametric ANCOVA

19. Secondary Outcome: Maximum Whole Blood Concentration (Cmax) for Bosentan and Its Metabolites, Ro 47-8634, Ro 48-5033, and Ro 64-1056 on Day 1
Description: Concentrations were measured directly in dried blood spot samples scheduled to be taken immediately prior to first study drug administration and at 0.5, 1, 2, 3, 7.5 and 12 hours post-dose on Day 1. Cmax was obtained directly from the measured concentrations. Cmax was corrected to a dose of 2 mg/kg bosentan (Cmaxc). The target dose was 2 mg/kg. However, as the smallest dose unit was 8 mg (quarter of a tablet), it was not possible to achieve the exact target dose in all patients. Therefore, Cmax was divided by the actual dose (in mg/kg) and multiplied by 2 mg/kg.
Time Frame: up to 12 hours
Population: Pharmacokinetic (PK) analysis set. This analysis set comprised all patients included in the all-treated set who were able to provide at least 5 of the 7 blood samples requested for at least one evaluable profile of PK assessment and who did not violate the protocol in a way that might affect the evaluation of the PK endpoints.
Measure: Geometric Mean (95% Confidence Interval); unit: ng/mL
Arm/Group | Bosentan
Number analyzed (Participants) | 11
ng/mL
  Bosentan | 30.1 [2.4 to 372.2]
  Ro 47-8634 | 0.1 [0.0 to 1.1]
  Ro 48-5033 | 0.6 [0.0 to 18.3]
  Ro 64-1056 | 0.9 [0.0 to 16.2]

20. Secondary Outcome: Cmax for Bosentan and Its Metabolites, Ro 47-8634, Ro 48-5033, and Ro 64-1056 on Day 5
Description: Concentrations were measured directly in dried blood spot samples scheduled to be taken immediately prior to study drug administration and at 0.5, 1, 2, 3, 7.5, and 12 hours post-dose on Day 5. Cmax obtained directly from the measured concentrations . Cmax was corrected to a dose of 2 mg/kg bosentan (Cmaxc). The target dose was 2 mg/kg. However, as the smallest dose unit was 8 mg (quarter of a tablet), it was not possible to achieve the exact target dose in all patients. Therefore, Cmax was divided by the actual dose (in mg/kg) and multiplied by 2 mg/kg.
Time Frame: 12 hours
Population: PK analysis set. This analysis set comprised all patients included in the all-treated set who were able to provide at least 5 of the 7 blood samples requested for at least one evaluable profile of PK assessment and who did not violate the protocol in a way that might affect the evaluation of the PK endpoints.
Measure: Geometric Mean (95% Confidence Interval); unit: ng/mL
Arm/Group | Bosentan
Number analyzed (Participants) | 7
ng/mL
  Bosentan | 880.0 [339.2 to 2282.7]
  Ro 47-8634 | 24.9 [9.0 to 69.1]
  Ro 48-5033 | 292.3 [115.8 to 738.1]
  Ro 64-1056 | 136.0 [77.4 to 238.8]

21. Secondary Outcome: Time to Maximum Whole Blood Concentration (Tmax) for Bosentan on Day 1
Description: Concentrations were measured directly in dried blood spot samples scheduled to be taken immediately prior to first study drug administration and at 0.5, 1, 2, 3, 7.5 and 12 hours post-dose on Day 1. Tmax was obtained directly from the measured concentrations.
Time Frame: up to 12 hours
Population: as for outcome 20
Measure: Median (Full Range); unit: hours
Arm/Group | Bosentan
Number analyzed (Participants) | 10
hours | 12.0 [7.5 to 12.0]

22. Secondary Outcome: Tmax for Ro 47-8634 on Day 1
Description: as for outcome 21
Time Frame: up to 12 hours
Population: as for outcome 20
Measure: Median (Full Range); unit: hours
Arm/Group | Bosentan
Number analyzed (Participants) | 5
hours | 12.0 [7.5 to 12.0]

23. Secondary Outcome: Tmax for Ro 48-5033 on Day 1
Description: as for outcome 21
Time Frame: up to 12 hours
Population: as for outcome 20
Measure: Median (Full Range); unit: hours
Arm/Group | Bosentan
Number analyzed (Participants) | 7
hours | 12.0 [12.0 to 12.0]

24. Secondary Outcome: Tmax for Ro 64-1056 on Day 1
Description: as for outcome 21
Time Frame: up to 12 hours
Population: as for outcome 20
Measure: Median (Full Range); unit: hours
Arm/Group | Bosentan
Number analyzed (Participants) | 8
hours | 12 [0.5 to 12.0]

25. Secondary Outcome: Tmax for Bosentan on Day 5
Description: Concentrations were measured directly in dried blood spot samples scheduled to be taken immediately prior to study drug administration and at 0.5, 1, 2, 3, 7.5, and 12 hours post-dose on Day 5. Tmax was obtained directly from the measured concentrations.
Time Frame: 12 hours
Population: as for outcome 20
Measure: Median (Full Range); unit: hours
Arm/Group | Bosentan
Number analyzed (Participants) | 7
hours | 7.5 [0.8 to 12.0]

26. Secondary Outcome: Tmax for Ro 47-8634 on Day 5
Description: as for outcome 25
Time Frame: 12 hours
Population: as for outcome 20
Measure: Median (Full Range); unit: hours
Arm/Group | Bosentan
Number analyzed (Participants) | 7
hours | 6.5 [0.8 to 12.0]

27. Secondary Outcome: Tmax for Ro 48-5033 on Day 5
Description: as for outcome 25
Time Frame: 12 hours
Population: as for outcome 20
Measure: Median (Full Range); unit: hours
Arm/Group | Bosentan
Number analyzed (Participants) | 7
hours | 7.5 [0.8 to 12.0]

28. Secondary Outcome: Tmax for Ro 64-1056 on Day 5
Description: as for outcome 25
Time Frame: 12 hours
Population: as for outcome 20
Measure: Median (Full Range); unit: hours
Arm/Group | Bosentan
Number analyzed (Participants) | 7
hours | 12.0 [7.5 to 12.0]

29. Secondary Outcome: Area Under the Concentration-time Curve Over a Period of 12 h (AUC0-12 Day 1)) for Bosentan and Its Metabolites, Ro 47-8634, Ro 48-5033, and Ro 64-1056 on Day 1
Description: Concentrations were measured directly in dried blood spot samples scheduled to be taken immediately prior to first study drug administration and at 0.5, 1, 2, 3, 7.5 and 12 hours post-dose on Day 1. Pharmacokinetic parameters were determined on the basis of scheduled blood sampling time points using non-compartmental analysis. Actual blood sampling times were used only if there was a deviation of more than 5% from the scheduled times. AUC0-12 Day 1 was calculated according to the trapezoidal rule using the measured concentration-time values above the limit of quantification.
Time Frame: 12 hours
Population: as for outcome 20
Measure: Geometric Mean (95% Confidence Interval); unit: h*ng/mL
Arm/Group | Bosentan
Number analyzed (Participants) | 11
h*ng/mL
  Bosentan | 163.9 [9.6 to 2795.4]
  Ro 47-8634 | 0.1 [0.0 to 3.7]
  Ro 48-5033 | 1.4 [0.0 to 69.9]
  Ro 64-1056 | 2.2 [0.1 to 64.1]

30. Secondary Outcome: Area Under the Concentration-time Curve Over a Dosing Interval at Steady State on Day 5 (AUCtau) for Bosentan and Its Metabolites, Ro 47-8634, Ro 48-5033, and Ro 64-1056
Description: Concentrations were measured directly in dried blood spot samples scheduled to be taken immediately prior to study drug administration and at 0.5, 1, 2, 3, 7.5, and 12 hours post-dose on Day 5. Pharmacokinetic parameters were determined on the basis of scheduled blood sampling time points using non-compartmental analysis. Actual blood sampling times were used only if there was a deviation of more than 5% from the scheduled times. AUCtau Day 5 was calculated according to the trapezoidal rule using the measured concentration-time values above the limit of quantification.
Time Frame: 5 days
Population: as for outcome 20
Measure: Geometric Mean (95% Confidence Interval); unit: h*ng/mL
Arm/Group | Bosentan
Number analyzed (Participants) | 7
h*ng/mL
  Bosentan | 6165.4 [2429.6 to 15645.3]
  Ro 47-8634 | 217.3 [75.3 to 626.8]
  Ro 48-5033 | 2839.5 [1155.2 to 6979.2]
  Ro 64-1056 | 1321.7 [729.5 to 2395.0]

31. Secondary Outcome: Area Under the Concentration-time Curve Over a Period of 24 h (Dose-corrected to 2 mg/kg) on Day 1 (AUC0-24C Day 1) for Bosentan and Its Metabolites, Ro 47-8634, Ro 48-5033, and Ro 64-1056
Description: Concentrations were measured directly in dried blood spot samples scheduled to be taken immediately prior to first study drug administration and at 0.5, 1, 2, 3, 7.5 and 12 hours post-dose on Day 1. Pharmacokinetic parameters were determined on the basis of scheduled blood sampling time points using non-compartmental analysis. Actual blood sampling times were used only if there was a deviation of more than 5% from the scheduled times. AUC0-24C Day 1 was calculated as a multiple of AUC0-12, (2 × AUC0-12 for 2 times daily dosing) corrected to 2 mg/kg.
Time Frame: 24 hours
Population: as for outcome 20
Measure: Geometric Mean (95% Confidence Interval); unit: h*ng/mL
Arm/Group | Bosentan
Number analyzed (Participants) | 11
h*ng/mL
  Bosentan | 287.5 [15.0 to 5504.7]
  Ro 47-8634 | 0.1 [0.0 to 6.1]
  Ro 48-5033 | 2.0 [0.0 to 125.8]
  Ro 64-1056 | 3.4 [0.1 to 120.8]

32. Secondary Outcome: Area Under the Concentration-time Curve Over a Period of 24 h (Dose-corrected to 2 mg/kg) on Day 5 (AUC0-24C Day 5) for Bosentan and Its Metabolites, Ro 47-8634, Ro 48-5033, and Ro 64-1056
Description: Concentrations were measured directly in dried blood spot samples scheduled to be taken immediately prior to study drug administration and at 0.5, 1, 2, 3, 7.5, and 12 hours post-dose on Day 5. Pharmacokinetic parameters were determined on the basis of scheduled blood sampling time points using non-compartmental analysis. Actual blood sampling times were used only if there was a deviation of more than 5% from the scheduled times. AUC0-24C Day 5 was calculated as a multiple of AUCtau, (2 × AUCtau for 2 times daily dosing) corrected to 2 mg/kg.
Time Frame: 24 hours
Population: as for outcome 20
Measure: Geometric Mean (95% Confidence Interval); unit: h*ng/mL
Arm/Group | Bosentan
Number analyzed (Participants) | 7
h*ng/mL
  Bosentan | 11530.2 [4507.0 to 29497.5]
  Ro 47-8634 | 406.3 [139.8 to 1180.9]
  Ro 48-5033 | 5310.3 [2184.4 to 12908.9]
  Ro 64-1056 | 2471.9 [1386.1 to 4408.0]

33. Secondary Outcome: Accumulation Index (AI) for Bosentan
Description: Concentrations were measured directly in dried blood spot samples scheduled to be taken immediately prior to first study drug administration and at 0.5, 1, 2, 3, 7.5 and 12 hours post-dose on Days 1 and 5. Pharmacokinetic parameters were determined on the basis of scheduled blood sampling time points using non-compartmental analysis. Actual blood sampling times were used only if there was a deviation of more than 5% from the scheduled times. AI was calculated as the ratio AUCtau /AUC0-12 for the subjects having PK samples collected on Day 1 and Day 5 and with AUC0-12 > 0 ng.h/mL.
Time Frame: 5 days
Population: as for outcome 20
Measure: Geometric Mean (95% Confidence Interval); unit: accumulation index
Arm/Group | Bosentan
Number analyzed (Participants) | 7
accumulation index | 61.6 [0.5 to 7813.9]

ADVERSE EVENTS:
Time Frame: Up to 21 Days, plus up to 60 days after end of treatment for serious adverse events
Arm/Group | Bosentan | Placebo
Serious Adverse Events (participants affected / at risk) | 2/13 | 3/8
Other Adverse Events (participants affected / at risk) | 9/13 | 2/8
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Bosentan (N=13) | Placebo (N=8)
HEPATITIS (Hepatobiliary disorders) | 1 | 0
METABOLIC ACIDOSIS (Metabolism and nutrition disorders) | 1 | 0
HYPERCAPNIA (Respiratory, thoracic and mediastinal disorders) | 1 | 0
PNEUMOTHORAX (Respiratory, thoracic and mediastinal disorders) | 0 | 2
CIRCULATORY COLLAPSE (Vascular disorders) | 1 | 0
SEPSIS (Infections and infestations) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Bosentan (N=13) | Placebo (N=8)
ANAEMIA (Blood and lymphatic system disorders) | 3 | 1
GENERALISED OEDEMA (General disorders) | 3 | 0
COAGULOPATHY (Blood and lymphatic system disorders) | 1 | 1
VOMITING (Gastrointestinal disorders) | 2 | 0
BILIRUBIN CONJUGATED INCREASED (Investigations) | 1 | 0
BODY TEMPERATURE INCREASED (Investigations) | 1 | 0
C-REACTIVE PROTEIN INCREASED (Investigations) | 1 | 0
DYSPHONIA (Respiratory, thoracic and mediastinal disorders) | 1 | 0
ENDOTRACHEAL INTUBATION COMPLICATION (Injury, poisoning and procedural complications) | 1 | 0
GASTRIC HAEMORRHAGE (Gastrointestinal disorders) | 1 | 0
HYPOGLYCAEMIA (Metabolism and nutrition disorders) | 0 | 1
HYPOKALAEMIA (Metabolism and nutrition disorders) | 0 | 1
HYPOPHOSPHATAEMIA (Metabolism and nutrition disorders) | 0 | 1
INFECTIOUS DISEASE CARRIER (Infections and infestations) | 1 | 0
METABOLIC ACIDOSIS (Metabolism and nutrition disorders) | 0 | 1
METHAEMOGLOBINAEMIA (Blood and lymphatic system disorders) | 1 | 0
MITRAL VALVE INCOMPETENCE (Cardiac disorders) | 1 | 0
PNEUMOMEDIASTINUM (Respiratory, thoracic and mediastinal disorders) | 1 | 0
PNEUMOTHORAX (Respiratory, thoracic and mediastinal disorders) | 1 | 0
PROCEDURAL COMPLICATION (Injury, poisoning and procedural complications) | 1 | 0
THROMBOCYTOPENIA (Blood and lymphatic system disorders) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other